CLINICAL TRIAL: NCT01337102
Title: Randomized Trial to Investigate the Impact of a Computer-Generated Quality of Life Assessment Program on Treatment Patterns for Advanced Non-Small Cell Lung Cancer Patients (LUNL2)
Brief Title: Computer-Generated Quality of Life Assessment Program for Advanced Non-Small Cell Lung Cancer Patients (LUNL2)
Acronym: LUNL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 04-0349-CE
Record Dates: First submitted 2011-04-05; First posted 2011-04-18 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Stage 3b; Stage 4; First Line Chemotherapy Treatment; Quality Of Life; Palliative Care; Randomized; Lung Cancer Scale
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physician to receive results (Other): Arm 1 Physician to receive the results of the Lung QoL scale
  Interventions: Procedure: Physician Receives QoL results
- Physician Does Not Receive Results (Other): Arm 2 Physician does not receive the results of the Lung QoL scale
  Interventions: Procedure: Physician Does not receive the results

INTERVENTIONS:
Procedure: Physician Receives QoL results — Patient completes the Lung Cancer QoL scale on the Palm held computer device and the Physician receives the print out of the results.
  Arms: Physician to receive results
Procedure: Physician Does not receive the results — Patient completes the Lung Cancer QoL scale on the Palm held computer device and the Physician does not receive the print out of the results.
  Arms: Physician Does Not Receive Results

SUMMARY:
In the treatment of advanced cancer, maximizing quality of life (QoL) is a fundamental goal for oncologists and their patients. In order to achieve this goal, some form of systematic and reliable QoL assessment is needed in routine clinical practice to evaluate the impact of advanced cancer treatments on QoL. The Lung Cancer Symptom Scale (LCSS) is a validated site-specific QoL measure designed for use in patients with lung cancer undergoing treatment. Recently it has been developed into an electronic form that uses a hand-held pocket personal computer (pc) to enhance collection and presentation of QoL assessments into clinical trials and patient care. This study will evaluate the impact of this computer-generated QoL (LCSS-QL) assessment on treatment practices for advanced lung cancer patients using a randomized trial design. The investigators hypothesize that a Computer-Generated Quality of Life Assessment Program will positively impact treatment patterns for patients with lung cancer.

Specifically, the investigators hypothesize:

1. Use of the LCSS-QL will increase and accelerate referral to and use of palliative care services;
2. Use of the LCSS-QL will decrease the duration of palliative chemotherapy treatment with earlier identification of lack of benefit in some patients;
3. Use of the LCSS-QL may decrease the use of imaging tests to assess objective tumor response as an indicator of treatment benefit.

Maximizing quality of life is one of the most important goals of palliative chemotherapy in the treatment of advanced lung cancer. If this simple practical tool can be demonstrated to improve palliative management of these patients, including optimizing duration of chemotherapy and use of palliative and supportive services based on patient QoL response, this will dramatically improve the quality of care provided to advanced lung cancer patients. This study will also provide a springboard for other ways to incorporate computer-generated QoL measurement in treatment decision-making in advanced cancer patients, including in other tumor types such as advanced breast and colorectal cancer.

DETAILED DESCRIPTION:
Study Design The study will be conducted using an unblinded, randomized trial design. Patients starting systemic therapy for advanced NSCLC will be invited to complete the LCSS-QL upon starting first-line systemic chemotherapy and then prior to subsequent treatment visits (every 3 weeks). Patients will then be randomized at baseline to whether or not their physician will receive this information at the time of clinic visits for the duration of study participation. Randomization codes will be generated by computer program, with stratification by physician, platinum-based versus non-platinum based therapy and Eastern Cooperative Group Performance Status 0 and 1 versus 2 and 3. All patients complete the LCSS-QL at baseline, at the beginning of each cycle of chemotherapy, and at follow up visits until disease progression (initiation of subsequent therapy)or discontinue clinic visits an expected average of 12 to 18 weeks.

Patient Population All NSCLC patients with advanced disease (Stage 3B or 4) starting systemic therapy at the Princess Margaret Hospital will be eligible to participate. Inclusion criteria include the physical ability to use the hand-held instrument (adequate vision, manual dexterity), provision of written informed consent, and written fluency in English, French, Italian, Spanish, Portuguese or Chinese. Patients will be excluded if they are unable to complete or understand the assessment process, or if they are receiving concurrent radical radiotherapy.

Physician Information Physicians will be trained in interpretation of the LCSS electronic output data, in order to facilitate interpretation of the different domains of patient well-being, for example pain scores. An endorsement sheet will be printed in addition to the LCSS data, highlighting major changes in quality of life. For example, deterioration in pain control will be highlighted with suggestions to increase or change pain medication, consider radiotherapy and other pain management options, including changing systemic therapy.

Outcomes

Endpoints include palliative care referral rates, duration of systemic therapy, use of supportive interventions and QoL during treatment.

Data on the number of chemotherapy cycles administered, referral to palliative care (including timing), institution of additional supportive treatments, and number of imaging tests ordered will be collected for all patients prospectively. Data on LCSS scores, subsequent therapy, and date of death will also be recorded.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of Primary Non Small Cell Lung Cancer
* Stage 3 or 4 Lung Cancer
* To receive 1st line Chemotherapy
* Platinum based chemotherapy or Non Platinum
* Physical ability to use the hand held device(adequate vision, manual dexterity),
* ECOG 1-2
* Written fluency in English, French, Italian, Spanish, Portuguese or Chinese

Exclusion Criteria:

* Patients will be excluded if they are unable to complete or understand the assessment process,
* If they are receiving concurrent radical radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2004-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of Palliative care Referrals. | Approximately 12 - 18 weeks
  To assess the impact of use of the LCSS-QL on palliative care referrals;
Number of palliative first-line chemotherapy cycles administered. | Approximately 12 - 18 weeks
  To assess the impact of use of the LCSS-QL on the number of palliative first-line chemotherapy cycles administered

SECONDARY OUTCOMES:
Use of supportive treatments. | 12 - 18 weeks
  To assess the impact of use of the LCSS-QL on the use of supportive treatments including radiotherapy, home oxygen, transfusion or growth factor support, community care support;
Number of imaging tests ordered. | Approximately 12 - 18 weeks
  To assess the impact of use of the LCSS-QL on the number of imaging tests ordered to evaluate patient response to therapy.
Differences between study arm scores | Approximately 12 - 18 weeks
  To compare LCSS-QL scores of patients between the two study arms

CONTACTS AND LOCATIONS:
Overall Officials: NATASHA LEIGHL, MD MSC, Principal Investigator — UNIVERSITY HEALTH NETWORK / PRINCESS MARGARET HOSPITAL
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada